CLINICAL TRIAL: NCT00286819
Title: Randomized Phase II Study of Dose-Dense Fluorouracil Plus Epirubicin 75 Plus Cyclophosphamide (FEC75) and Fluorouracil Plus Epirubicin 90 Plus Cyclophosphamide (FEC90) as Adjuvant Therapy for Early Breast Cancer
Brief Title: Dose Density FU 75 and FU 90 as Adjuvant Therapy for Early Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Central European Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CECOG/Breast.2.2.005
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer
Keywords: early breast cancer,; Fluorouracil
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- the FEC75 regimen (Experimental): Arm A: the FEC75 regimen will be given at the following doses:
  Fluorouracil 500mg/m2 by i.v. bolus or infusion. Epirubicin 75mg/m2 by 30 minutes i.v infusion and Cyclophosphamide 500mg/m2 by i.v bolus or infusion. All three drugs will be administered intravenously on Day 1 of each 14-day cycles.
  Interventions: Drug: the FEC75 and 95 regimen
- FEC90 regimen (Experimental): Arm B: the FEC90 regimen will be given at the following doses:
  Fluorouracil 500mg/m2 by i.v. bolus or infusion.Epirubicin 90mg/m2 by 30 minutes i.v infusion and Cyclophosphamide 500mg/m2 by i.v bolus or infusion.
  All three drugs will be administered intravenously on Day 1 of each 14-day cycles.
  Pegfilgrastim fixed dose of 6mg as a single subcutaneous injection will be given in both arms on Day 2 of each cycle.
  Interventions: Drug: the FEC75 and 95 regimen

INTERVENTIONS:
Drug: the FEC75 and 95 regimen — Fluorouracil 500mg/m2 by i.v. bolus or infusion. Epirubicin 75mg/m2 by 30 minutes i.v infusion and Cyclophosphamide 500mg/m2 by i.v bolus or infusion. All three drugs will be administered intravenously on Day 1 of each 14-day cycles.
  Arm B: the FEC90 regimen will be given at the following doses:
  Fluorouracil 500mg/m2 by i.v. bolus or infusion.Epirubicin 90mg/m2 by 30 minutes i.v infusion and Cyclophosphamide 500mg/m2 by i.v bolus or infusion.
  All three drugs will be administered intravenously on Day 1 of each 14-day cycles.
  Pegfilgrastim fixed dose of 6mg as a single subcutaneous injection will be given in both arms on Day 2 of each cycle.
  Six cycles of adjuvant chemotherapy will be administered in both arms (A + B

SUMMARY:
This is an open -label randomized phase II study of dose-dense Fluorouracil/Epirubicin/Cyclophosphamide (FEC) administered with Epirubicin of 75mg/m2 (FEC75) and Epirubicin 90mg/m2 (FEC90) in untreated patients with early breast cancer.

DETAILED DESCRIPTION:
Arm A: the FEC75 regimen will be given at the following doses:

Fluorouracil 500mg/m2 by i.v. bolus or infusion. Epirubicin 75mg/m2 by 30 minutes i.v infusion and Cyclophosphamide 500mg/m2 by i.v bolus or infusion. All three drugs will be administered intravenously on Day 1 of each 14-day cycles.

Arm B: the FEC90 regimen will be given at the following doses:

Fluorouracil 500mg/m2 by i.v. bolus or infusion.Epirubicin 90mg/m2 by 30 minutes i.v infusion and Cyclophosphamide 500mg/m2 by i.v bolus or infusion.

All three drugs will be administered intravenously on Day 1 of each 14-day cycles.

Pegfilgrastim fixed dose of 6mg as a single subcutaneous injection will be given in both arms on Day 2 of each cycle.

Six cycles of adjuvant chemotherapy will be administered in both arms (A + B)

ELIGIBILITY:
Inclusion Criteria:

* patients with histological diagnosis of invasive breast cancer
* Patients with early stage I, II,III breast cancer amendable for complete surgical resection.
* Patients with any nodal status
* Patients with ER and PR -negative tumors. In case of axillary involvement:any hormonal receptors status.
* perfomance Status 0-1 on the ECOG Scale
* patients indicated for adjuvant chemotherapy
* No previous chemotherapy or radiotherapy
* Patients have to be randomized within 8 weeks after surgery. Its recommended that patients will start chemotherapy within 1 month after surgical treatment.

Exclusion Criteria:

* active infection
* pregnancy/breast feeding
* serious concomitant systemic disorders incompatible with the study
* Second primary malignancy (expect in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin)
* Use of any other investigational agent within 4 weeks before enrollment into the study
* Cocurrent administration of radiation therapy, chemotherapy, hormonal therapy or immunotherapy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-04; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
The primary objective of this randomized phase II is to determine the relative dose intensity (RDI) of six adjuvant cycles of FEC75 and FEC90 regimens given every 14 days with pegfilgrastim (Neulasta) support in subjects with early breast cancer.

SECONDARY OUTCOMES:
- Incidence of dose delays and dose reductions of planned chemotherapy due to neutropenic events
-Toxicity and tolerability
-disease Free survival (As neither radiotherapy nor hormone therapy are specified and will be carried out according to institutional guidelines, DST has t be interpreted with caution)
- Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Brodowicz, Prof, Principal Investigator — Univ. Klinik für innere Medizin I
Locations (5):
- AKH, Universitätsklinik für Innere Medizin 1, Vienna, Austria
- Onkotherápiás Klinika,, Szeged, Hungary
- Medical University of Gdansk, Dept. of Oncology and Radiotherapy, Gdansk, Poland
- Slovakia (2):
  - Nomocnica Sv. Alzbety, Narodny Onkologicky Ustav, Bratislava
  - Oncology Institute, Department of Radiotherapy and Onclogy, Košice